CLINICAL TRIAL: NCT04277507
Title: A Prospective, Multicenter Study of the AERin Medical Vivaer® ARC Stylus for Nasal AirWAY Obstruction (AERWAY)
Brief Title: Study of the AERin Medical Vivaer® ARC Stylus for Nasal AirWAY Obstruction
Acronym: AERWAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aerin Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP900
Record Dates: First submitted 2020-02-17; First posted 2020-02-20 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Nasal Obstruction
Keywords: Nasal valve; Nasal airway obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Vivaer Stylus (Experimental): Intervention: Procedure: thermal treatment of submucosal tissue including cartilage in the internal nasal valve area
  Interventions: Device: Vivaer Stylus

INTERVENTIONS:
Device: Vivaer Stylus — Delivery of low-power, temperature-controlled, radiofrequency energy to the tissues of the internal nasal valve area
  Other Names: Aerin Medical Device

SUMMARY:
Post-market study to continue to evaluate the effectiveness of the Vivaer® ARC Stylus for nasal airway obstruction

DETAILED DESCRIPTION:
Prospective, Multicenter, Non-randomized Study of the Aerin Medical Vivaer® ARC Stylus for Nasal Airway Obstruction to continue to evaluate the effectiveness of the Vivaer® ARC Stylus for treating the nasal valve area to improve symptoms in those diagnosed with nasal airway obstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Willing and able to provide informed consent
3. Willing and able to comply with the study protocol
4. Seeking treatment for nasal obstruction
5. NOSE score of ≥ 60 at Baseline
6. Nasal valve is a primary or significant contributor to the subject's nasal obstruction as determined by the study investigator (based on clinical presentation, physical examination, nasal endoscopy, etc.) and the subject has a positive response to any of the following temporary measures (based on patient history or office exam):

   * Use of external nasal dilator strips (e.g., Breathe Right Strips)
   * Q-Tip test (manual intranasal lateralization)
   * Use of nasal stents
   * Cottle Maneuver (manual lateral retraction of the cheek)

Exclusion Criteria:

1. Prior surgical treatment of the nasal valve
2. Rhinoplasty, septoplasty, inferior turbinate reduction or other surgical nasal procedures within the past three (3) months
3. Anatomy that requires an adjunctive surgical nasal procedure on the same day or 3 months after the Vivaer procedure
4. Medical conditions which in the opinion of the treating physician would predispose the subject to poor wound healing or increased surgical risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2024-10-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Alabama Nasal and Sinus Center, Birmingham, Alabama
  - Arizona Desert ENT Specialists, Goodyear, Arizona
  - Sacramento ENT, Roseville, California
  - ENT Associates of South Florida, Boca Raton, Florida
  - ENT Associates of South Florida, Plantation, Florida
  - Chicago Nasal and Sinus Center, Chicago, Illinois
  - Baton Rouge General / Sinus and Nasal Specialists of Louisiana, Baton Rouge, Louisiana
  - Advocare Aroesty ENT Associates, Mount Arlington, New Jersey
  - UT Physicians Otorhinolaryngology - Texas Medical Center, Houston, Texas
  - ENT Associates of Texas, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yao WC, Pritikin J, Sillers MJ, Barham HP. Two-year outcomes of temperature-controlled radiofrequency device treatment of the nasal valve for patients with nasal airway obstruction. Laryngoscope Investig Otolaryngol. 2023 Jun 15;8(4):808-815. doi: 10.1002/lio2.1089. eCollection 2023 Aug. PMID 37621275
- [Result] Yao WC, Ow RA, Barham HP (2021) Temperature-Controlled Radiofrequency Treatment of the Nasal Valve and Nasal Airway Obstruction: Early Results of a Prospective, Multi-Center Study. J Otolaryngol Rhinol 7:104. doi.org/10.23937/2572-4193.1510105
- [Result] Yao WC, Ow R, Sillers MJ, Nachlas NE, Johnson CD, Ehmer D, Pritikin J, Barham HP. Three-Year Outcomes After Temperature-Controlled Radiofrequency Treatment of Nasal Airway Obstruction. OTO Open. 2025 Apr 7;9(2):e70111. doi: 10.1002/oto2.70111. eCollection 2025 Apr-Jun. PMID 40196218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment was "Up to 125 treated patients" to be enrolled in the study at up to 20 sites (medical clinics) in the United States. Recruitment occurred 01FEB2020 - 26AUG2020.
Groups:
- Vivaer Treatment: Single Arm Study. Eligible subjects who have signed consent and qualify will have their nasal valve treated in a single Vivaer® treatment session and will be considered enrolled once the device has entered the nasal cavity.
Period: Overall Study
Arm/Group | Vivaer Treatment
Started | 122
Completed | 91 (A total of 122 patients were treated and 91 reached (24M Visit) 2 years. The study is still in follow-up through 36M (3 years).)
Not Completed | 31
Not completed — Lost to Follow-up | 17
Not completed — Completed through 24M but not interested in extension to 36M | 3
Not completed — Received Treatment Outside of Study that could affect study results | 2
Not completed — Withdrawal by Subject | 3
Not completed — Death due to COVID-19 | 1
Not completed — Data missing for full evaluation | 5

BASELINE CHARACTERISTICS:
Groups:
- Vivaer Treatment: Intervention: Procedure: thermal treatment of submucosal tissue including cartilage in the internal nasal valve area
  Vivaer Stylus: Delivery of low-power, temperature-controlled, radiofrequency energy to the tissues of the internal nasal valve area
Arm/Group | Vivaer Treatment
Number analyzed (Participants) | 122
Age, Customized [Count of Participants; unit: Participants]
  <60 years | 83
  >=60 years | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 107
  Black or African American | 4
  Asian | 3
  Asian, White | 2
  Black or African American, White | 1
  Declined Available Choices | 5
Baseline NOSE Scale Score [Mean (Standard Deviation); unit: units on a scale] — Nasal Obstruction Symptom Evaluation Scale (NOSE scale). Subject completed 1 month review of the following 5 categories: Nasal Congestion/Stuffiness; Nasal Blockage or Obstruction; Trouble Breathing through my nose; Trouble Sleeping/ Unable to get enough air through my nose during exercise or exertion. Subjects answer 0-4 (0=not a problem; 1=very mild problem; 2=moderate problem; 3fairly bad problem; 4=severe problem) answers are multiplied by 5, score is out of 100
  units on a scale | 80.3 (12.6)
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] — Average Body Mass Index across all subjects
  Kg/m^2 | 27.6 (6.7)
Nasal Valve Collapse Mechanism [Count of Participants; unit: Participants]
  Bilateral Dynamic | 68
  Bilateral Static | 47
  Unilateral Dynamic | 2
  Unilateral Dynamic and Unilateral Static | 2
  Unilateral Static | 1
  Unreported | 2
Additional Nasal Obstruction Diagnosis [Count of Participants; unit: Participants]
  Nasal Valve Stenosis | 64
  Septal Turbinate (Nasal Septal Body) | 37
  Septal Deviation | 34
  Turbinate Enlargement | 31
  Nasal Polyps | 3
History of Nasal Surgery [Count of Participants; unit: Participants] | 67

OUTCOME MEASURES:

1. Primary Outcome: Change in Nasal Obstructive Symptom Evaluation (NOSE) Scores From Baseline to 3 Months
Description: Mean change in NOSE score from Baseline to 3 months.Scores may range from the best score of 0, meaning no nasal obstructive symptoms to the worst score of 100, meaning severe nasal obstructive symptoms.
Time Frame: 3 Month
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Protocol Eligible Subjects: Scores per-protocol eligible subjects total 119 at 3M
Arm/Group | Protocol Eligible Subjects
Number analyzed (Participants) | 119
score on a scale | -47.6 (26.1)

2. Other Pre Specified Outcome: Subject-reported Visual Analog Scale (VAS) Pain Scores in Relation to the Area Treated by the Study Procedure
Description: The Pain VAS will be used to rate pain associated with the treatment (Hawker, Mian et al. 2011). Subjects are asked to mark their pain level on a 10 cm line anchored by verbal descriptors: 0 = no pain and 10 = worst pain imaginable. The study staff will measure with a metric ruler from the 0, the beginning of the line, to the vertical mark made by the subject. The result, expressed in millimeters, will represent the subject's VAS Pain Score with 100 being the worst pain imaginable.
Time Frame: 3 months post study procedure
Population: All treated subjects VAS score at 3 months post procedure
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Vivaer Treatment
Number analyzed (Participants) | 122
millimeters | 4.5 (8.8)

3. Other Pre Specified Outcome: Subject Reported Change in Medication Use for Nasal Obstruction Symptoms
Description: Evaluate change (reduction) in medication used for nasal obstruction symptoms from Baseline to follow up timepoints post study procedure of 3 months, 6 months, 12 months and 24 months
Time Frame: 24 Month
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Taking Oral Medications at Baseline for NAO Symptoms: Subjects using Oral Medications at baseline for the relief of NAO Symptoms
- Subjects Using Nasal Sprays for NAO Symptoms: Subject using nasal sprays at baseline for the relief of NAO symptoms
Arm/Group | Subjects Taking Oral Medications at Baseline for NAO Symptoms | Subjects Using Nasal Sprays for NAO Symptoms
Number analyzed (Participants) | 63 | 66
Participants | 31 | 34

4. Other Pre Specified Outcome: Change in Nasal Obstructive Symptom Evaluation (NOSE)Scores From Baseline to 24 Months - Analysis
Description: Mean change in NOSE score from Baseline to 24 months post study procedure. Scores may range from the best score of 0, meaning no nasal obstructive symptoms to the worst score of 100, meaning sever nasal obstructive symptoms
Time Frame: 24 Months
Population: A total of 1010 patients reached 2 year follow-up, of which, 12 had an additional nasal procedure and were reviewed separately
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Analysis Cohort (24)M (Vivaer Treatment): 89 Eligible subjects who completed through 24 month visit with 12 excluded for anyaisis
Arm/Group | Analysis Cohort (24)M (Vivaer Treatment)
Number analyzed (Participants) | 89
score on a scale | 57 (2.8213)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Vivaer Treatment
All-Cause Mortality (participants affected / at risk) | 1/122
Serious Adverse Events (participants affected / at risk) | 1/122
Other Adverse Events (participants affected / at risk) | 0/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivaer Treatment (N=122)
Events Leading to Death (Infections and infestations) | 1 (1) — COVID-19
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — Severe Abdominal Pain
Corneal Damage (Eye disorders) | 1 (1)
Worsening Nasal Airway Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Psychiatric Disorder (Psychiatric disorders) | 1 (2)
Ankle Break (Musculoskeletal and connective tissue disorders) | 1 (1)
pulmonary Alveolar Protenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 1 (1)
Aortic Stenosis (Cardiac disorders) | 1 (1)
Ischemic Attack (Nervous system disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of this study are its lack of a control arm and the non-blinded nature of this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT04277507/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT04277507/SAP_001.pdf
  • Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT04277507/ICF_002.pdf